CLINICAL TRIAL: NCT05463029
Title: Advanced Resting State fMRI for Clinical Evaluation of Brain Network Integrity in Disorders of Consciousness
Brief Title: Resting State fMRI in Disorders of Consciousness
Status: Terminated | Type: Observational
Why Stopped: This protocol was merged into another study
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jeffery Ware, Medical Doctor, University of Pennsylvania
Other Study IDs: 851120
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Disorders of Consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Healthy control participants will be recruited from the general population through the use of flyers and other means of advertising.
- Affected Patients: Research staff locate eligible patients in the hospital through real-time medical record review at the time of initial presentation to the NICU or request for neurology consultation for patients in the MICU or CCU. Once potential patients have been identified, research staff will approach their Legally Authorized Representative to introduce the study and initiate the informed consent process, if appropriate.

SUMMARY:
Disorders of consciousness (DoC) remain a major clinical challenge in which high rates of misdiagnosis and difficult prognostication stem from limitations in the ability to access the disordered physiological processes mechanisms of coma in real world clinical settings. There is a great need to develop, validate, and translate to clinical use reliable diagnostics to detect brain recovery potential not evident on neurobehavioral assessment. While resting state fMRI (rs-fMRI) has demonstrated potential to improve the diagnostic evaluation of DoC by detecting features of consciousness that are occult at bedside evaluation, this technology has yet to achieve widespread clinical utility. The investigators propose that recent advancements in rs-fMRI capabilities can be combined with streamlined analysis and interpretation approaches to overcome persistent intensive care unit to perform rs-fMRI in patients with prolonged impaired consciousness due to several causes including TBI, cardiac arrest, stroke, seizures, and severe CNS infection. The investigators will determine the optimal methods of data acquisition, analysis and interpretation for predicting recovery of consciousness in these patients. Our expectations are that this approach will produce highly reliable functional connectomic characterization of individual DoC patients, thereby allowing for more accurate outcome prediction. The investigators will additionally investigate the utility of a novel, simplified radiological approach to rs-fMRI data interpretation in comparison to computationally intensive connectomic approaches. This exploratory/developmental project is expected to provide critical data needed to design and appropriately power future R01 studies validating the efficacy of fMRI-based network integrity in the clinical evaluation of DoC.

DETAILED DESCRIPTION:
Disorders of consciousness (DoC) are states of altered consciousness stemming from an acquired injury to brain networks regulating arousal and awareness, characterized by a loss of excitatory neural activity across corticocortical, thalamocortical and thalamostriatal connections. DoC may be due to several causes including traumatic brain injury, anoxic brain injury from cardiac arrest, stroke, severe brain infections, prolonged seizures, or others. A primary challenge in the clinical management of DoC is accurately determining the type of DoC and level of consciousness, as well as the potential for recovery. This is crucial for decision-making and clinical management, with misdiagnosis rates as high as 40% due to limitations of clinical evaluation. Recent research has demonstrated that consciousness not detectable at bedside evaluation may be present in as many as 15-20% patients with DoC. Thus, to improve the clinical assessment of DoC and ultimately develop targeted interventions to promote neurological recovery, better methods of assessing DoC in individual patients must be developed, validated, and translated to clinical use. The use of rs-fMRI in the study of DoC has led to important insights into the biological mechanisms of coma as well as recovery of consciousness, yet the translation of rs-fMRI to the clinical management of individual patients with impaired consciousness has been hampered by several factors. First, BOLD fMRI reflects a complex combination of signals derived not only from neural activity but also from non-neurological sources that ultimately comprise as much as 25% of the BOLD signal obscuring true neural connectivity and introducing spurious connectivity. This limitation has usually been circumvented by analyzing fMRI at the group level, leveraging the statistical benefits of averaging data across individuals. Better strategies to distinguish between neural and non-neural contributors to the BOLD signal are needed to translate rs-fMRI to clinical use in individual patients. Additionally, conventional acquisition and analysis strategies have generally been shown to produce reliable estimates of functional connectivity only at clinically intractable scan times. Recent evidence suggests that highly reliable measures of functional connectivity can be obtained at the individual level at clinically feasible scan times using more advanced imaging protocols, outperforming even several-fold longer conventional acquisitions. The measured BOLD signal can be represented as a function of the signal intensity at excitation (S0), the echo time, and signal decay constant. Neural activity affects the BOLD signal by inducing an increase in blood-flow, which reduces the local concentration of deoxyhemoglobin and in turn decreases the local magnetic susceptibility thereby reducing the rate of transverse magnetization decay. By examining the signal decay across multiple echo times, changes in T2* can be distinguished from changes in S0 thereby allowing neural and non-neural signals from BOLD data to be differentiated. With sensitivity to BOLD signal being maximal near the T2*, multi-echo acquisitions can also enhance BOLD sensitivity by placing greater weight on those echoes closest to the T2* of a particular voxel ("optimally combining"), which is known to vary across the brain. Lastly, the process of combining BOLD data across echoes carries the advantage of dampening thermal noise which is randomly organized and tend to cancel out upon averaging. When combined with additional strategies to remove global motion-related signals, the influence of motion on BOLD data can be nearly eliminated. Only recently with the integration of other technical advances such as simultaneous multi-slice has it become possible to acquire multi-echo rs-fMRI without major compromises in spatial or temporal resolution acquisition. Practical challenges to obtaining advanced MRI in critically ill patients include the need to transport patients to research MRI instrumentation capable of the latest acquisition methods that have traditionally been located on different floors or even different buildings than intensive care units (ICUs). As a result, advanced MRI methods such as multi-echo rs-fMRI have mainly been applied to healthy subjects. This project will take advantage of a newly installed research-dedicated state-of-the-art 3 Tesla MRI system equipped with fast gradients a 32-channel receiver array embedded within the neurointensive care unit (NICU). This system is capable of multi-echo rs-fMRI at high spatiotemporal resolution and a key goal of this project is to determine whether functional network integrity in patients with DoC can be more reliably detected using multi-echo rs-fMRI than with standard rs-fMRI. Optimal methods would be unsupervised, capable of accommodating interindividual differences in functional topology, and capable of reducing complex connectivity data to discrete, clinically actionable insights. Another key goal of this project is to compare three approaches to connectome construction and characterization in their reliability at the individual patient level and degree of association with clinical measures of neurologic dysfunction and outcome. The first and most traditional approach will rely upon transformation of each data to a template space and node definition based upon group-level meta- analysis. The second approach will use a previously-described method of subject-level parcellation based upon connectivity gradients and ultimately compared across individuals based upon the degree of similarity to template networks. The final approach will use a radiological interpretation scheme in which expert neuroimagers trained to recognize typical spatial patterns of resting state networks will render an interpretation of the degree network maps obtained from independent component analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older diagnosed with acute DoC (defined by a Glasgow Coma Scale (GCS) motor score less than 6 and GCS verbal score less than 3 persisting at least 48 hours) due to trauma, cardiac arrest, stroke, seizure, or severe CNS infection.

Exclusion Criteria:

* Children under 18
* Contraindications to MRI (medical instability, non-MRI compatible implanted devices, retained metallic foreign bodies, claustrophobia)
* Presence of artifact-producing intracranial devices (aneurysm clips/coils, ventricular drains, craniectomy mesh, etc.)
* Large space-occupying lesions (50 mL) or substantial mass effect (herniation, 5mm midline shift) on preceding brain imaging
* Imminently life-threatening co-morbid conditions
* History of premorbid disabling neurological or psychiatric disease
* Current substance abuse or remote substance abuse with permanent organic sequelae
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with prolonged impaired consciousness (greater than 48 hours) due to several causes including TBI, cardiac arrest, stroke, seizures, and severe CNS infection. Demographically-similar healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Interclass correlation coefficient of functional-connectivity measures | Assessed at the time of the scan (for the coma patients within 1 week of DoC onset).
  The interclass correlation coefficient (ICC) is used to assess the reliability of functional connectivity measures.

SECONDARY OUTCOMES:
Glasgow Coma Scale (GCS) | The GCS is assessed at the time of the scan as well as at 10 days post-MRI.
  Ordinal scale describing the level of consciousness in a brain-injured patient.
Physical therapy-based functional status examination scores | Physical therapy-based functional status exam scores are assessed at 10 days post-MRI
  Measures of functional status scored on the Coma Recovery Scale-Revised (CRS-R) on a scale of 0-23 with a higher score indicating better function.
Weighted Kappa of radiological connectivity ratings | Assessed at the time of the scan (for the coma patients within 1 week of DoC onset).
  Used to assess the inter-rater reliability of radiological connectivity assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Ware, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT05463029/ICF_000.pdf